CLINICAL TRIAL: NCT02888821
Title: School-Home Program for Mexican Children With Attention and Behavioral Concerns
Acronym: CLS-FUERTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-19845
Record Dates: First submitted 2016-08-09; First posted 2016-09-05 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLS-FUERTE (Experimental): Families will receive the CLS-FUERTE intervention in the fall of the 2016-2017 school year. CLS-FUERTE includes caretaker, child and teacher components implemented during a 6 week period. All content of group sessions will be derived from the manualized CLS-FUERTE treatment protocol developed by the PI and study staff.
  Interventions: Behavioral: CLS-FUERTE
- Business as Usual (BAU) Waitlist Control (Other): Families will receive school services as usual while on a waitlist to receive CLS-FUERTE in the spring of the 2016-2017 school year.
  Interventions: Behavioral: CLS-FUERTE

INTERVENTIONS:
Behavioral: CLS-FUERTE — The CLS-FUERTE program is an approximately 6-week program and includes school (behavioral consultation with teachers), caretaker (caretaker skills groups), and student (skills groups) components which are integrated via joint teacher, parent, and student meetings and use of integrated behavioral programs in the classroom, on the playground, and at home.

SUMMARY:
A school-based behavioral intervention for Mexican youth with attention/behavior concerns (the Collaborative Life Skills Program for Latinos/Familias Unidades Empezando Retos y Tareas para el Éxito [CLS-FUERTE]:) will be pilot-tested in a mixed-method investigation with four Mexican elementary schools.

DETAILED DESCRIPTION:
A school-based behavioral intervention for Mexican youth with attention/behavior concerns (the Collaborative Life Skills Program for Latinos/Familias Unidades Empezando Retos y Tareas para el Éxito [CLS-FUERTE]:) will be pilot-tested in a mixed-method investigation with four Mexican elementary schools.

Participants will include 24-32 students (n = 6-8 per 4 schools) in participating schools. School personnel will help identify students with and at-risk for Attention-Deficit/Hyperactivity Disorder (ADHD) with at least one caretaker and teacher able to participate in the intervention. Students must be in 1st-6th grade at a participating school and must demonstrate clinically significant attention/behavioral concerns and related impairment as rated by caretakers and teachers. Caretakers and teachers must be able to attend program sessions held at the child's school over an approximately 6-week period. Through a school-clustered random assignment design, two schools will be selected to receive CLS-FUERTE during the fall of the 2016-2017 school year and two schools will be selected to receive school services as usual while waiting to receive CLS-FUERTE the spring of the 2016-2017 school year. Caregivers and teachers of students will complete questionnaires about child behavior and family functioning and caregivers will participate in focus groups at 4 time points regardless of treatment assignment: Pre (prior to random assignment), Post 1 (following CLS-FUERTE in the fall cohort), Post 2 (following CLS-FUERTE for in spring cohort), and Follow-up (at the end of the school year).

Feasibility and acceptability of CLS-FUERTE will be examined via participation enrollment, attendance, and engagement ratings and focus group feedback. Improvement in satisfaction with school services and youth outcomes will be examined and estimates of effect sizes will be used to support future scaled-up investigation.

ELIGIBILITY:
Inclusion Criteria:

* Caretakers and teachers of children must each describe at least 3 symptoms of ADHD as occurring "often" or "very often," as well as 1 impairment domain of ADHD as affecting the child "quite a bit" or "a lot" on a symptom screening interview.

Exclusion Criteria:

* Inability of caretakers or teachers to attend groups and meetings.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
ADHD Symptoms Change | Change in ADHD symptoms measured 3 times (i.e., from baseline at 3, 6, and 8 months)
  via parent and teacher rated questionnaire (i.e., the Child Symptom InventCLS-FUERTE completion), and Time 4 (end of the school year).
ADHD Impairment Change | measured 3 times (i.e., from baseline at 3, 6, and 8 months)
  via parent and teacher rated questionnaire (i.e., the Impairment Rating Scale [IRS] by Fabiano et al., 2006; the ADHD-FX by Haack et al., 2014; and the FX-II by Haack et al., unpublished).

SECONDARY OUTCOMES:
Executive Functioning Change | Change measured 3 times (i.e., from baseline at 3, 6, and 8 months)
  via parent and teacher rated questionnaire (i.e., the Behavior Rating Inventory of Executive Functioning-2 [BRIEF] by Gioia et al., 2000).

REFERENCES:
- See also: original CLS intervention efficacy study — http://dx.doi.org/10.1016/j.jaac.2016.05.023

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT02888821/Prot_SAP_000.pdf